CLINICAL TRIAL: NCT00092534
Title: A Randomized, Worldwide, Placebo-Controlled, Double-Blind Study to Investigate the Safety, Immunogenicity, and Efficacy on the Incidence of HPV 16/18-Related CIN 2/3 or Worse of the Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in 16- to 23-Year Old Women - The FUTURE II Study (Females United to Unilaterally Reduce Endo/Ectocervical Disease)
Brief Title: Cervical Intraepithelial Neoplasm (CIN) in Women (Gardasil) (V501-015)
Acronym: FUTURE II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: V501-015; 2004_082; V501-015 (Other: MSD)
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Genital Warts
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Vaccines, Synthetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadrivalent Human Papillomavirus (HPV) Vaccine (Experimental): The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 1 were vaccinated (at Day 1, Month 2 and Month 6) with the Quadrivalent HPV vaccine.
  Interventions: Biological: Gardasil, human papillomavirus (type 6, 11, 16, 18) recombinant vaccine
- Placebo (Placebo Comparator): The Vaccination Period for the base study encompassed Day 1 through Month 7, during which time study subjects in Group 2 were vaccinated (at Day 1, Month 2 and Month 6) with placebo.
  Interventions: Biological: Matching Placebo

INTERVENTIONS:
Biological: Gardasil, human papillomavirus (type 6, 11, 16, 18) recombinant vaccine — A 0.5 mL intramuscular injection in the deltoid muscle at Day 1, Month 2, and Month 6 in the Base Study.
  Other Names: V501, qHPV vaccine
  Arms: Quadrivalent Human Papillomavirus (HPV) Vaccine
Biological: Matching Placebo — A placebo 0.5 mL intramuscular injection in the deltoid muscle at Day 1, Month 2, and Month 6 in the Base Study.
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to determine if GARDASIL™ (V501) is able to prevent cervical cancer.

DETAILED DESCRIPTION:
In the 4-year Base Study (V501-015) (NCT00092534), participants were randomized in a 1:1 order to receive 3 doses of GARDASIL™ or matching placebo at Day 1, Month 2, and Month 6 and were assessed for efficacy, immunogenicity, and safety.

In the Base Study Extension (EXT) [V501-015-10], participants who received placebo or only 1 dose of GARDASIL™ in the Base Study, were given 3 doses of open-label GARDASIL™ at EXT Day 1, EXT Month 2, and EXT Month 6, and were followed to EXT Month 7. Participants who who received 2 doses of GARDASIL™ in the Base Study were given 1 dose of GARDASIL™ at EXT Day 1 and were followed for 15 days (day of vaccination plus 14 days).

In the 10-year Base Study Long-Term Follow-Up (LTFU) [V501-015-21] the effectiveness, immunogenicity and safety of GARDASIL™ was assessed during a period of 10 years following completion of the Base Study (V501-015) [14 years after the first dose of GARDASIL™] and, for some measures, the Base Study EXT (V501-015-10) [10 years after the first dose of GARDASIL™]. Participants from Denmark, Iceland, Norway and Sweden who participated in the Base Study were eligible to enroll in the LTFU. Effectiveness and safety was assessed by registry-based follow-up, and immunogenicity was assessed by serological testing at approximately Year 5 and Year 10 of the V501-015-21 LTFU.

An 8-year extension was added to the LTFU (V501-015-22] to continue the evaluation of the long-term effectiveness and immunogenicity of GARDASIL™. Effectiveness and safety will be assessed by registry-based follow-up, and immunogenicity will be assessed by serological testing at approximately Year 4 and Year 8 of the extension of the LTFU.

ELIGIBILITY:
Inclusion Criteria for the Base Study:

* Healthy women with an intact uterus with lifetime history of 0-4 sexual partners

  --For Extension Phase:
* Participant received placebo or an incomplete vaccination series in the original study

  --For LTFU:
* Participant was randomized into the Base Study from Denmark, Iceland, Norway, or Sweden.
* Agreed to allow passive follow-up (retrospective review of registry data), analysis of biopsy specimens, future contact from National Registry Study Center and serum collection

Exclusion Criteria for the Base Study:

* Prior Human Papilloma Virus (HPV) vaccination
* Prior abnormal Paps
* Prior history of genital warts

  --For Extension Phase:
* Prior complete HPV vaccination series
* Subject lives in a country in which Gardasil is approved and is within the age range of the local labeling for Gardasil

  --For LTFU Study:
* There were no exclusion criteria that did not overlap the inclusion criteria for this study.

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12167 (Actual)
Dates: Start 2002-06-14 (Actual); Primary Completion 2007-07-31 (Actual); Study Completion 2025-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Garland SM, Steben M, Sings HL, James M, Lu S, Railkar R, Barr E, Haupt RM, Joura EA. Natural history of genital warts: analysis of the placebo arm of 2 randomized phase III trials of a quadrivalent human papillomavirus (types 6, 11, 16, and 18) vaccine. J Infect Dis. 2009 Mar 15;199(6):805-14. doi: 10.1086/597071. PMID 19199546
- [Background] Barr E, Gause CK, Bautista OM, Railkar RA, Lupinacci LC, Insinga RP, Sings HL, Haupt RM. Impact of a prophylactic quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like particle vaccine in a sexually active population of North American women. Am J Obstet Gynecol. 2008 Mar;198(3):261.e1-11. doi: 10.1016/j.ajog.2007.09.001. PMID 18313445
- [Background] Joura EA, Leodolter S, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Garland SM, Harper DM, Tang GW, Ferris DG, Steben M, Jones RW, Bryan J, Taddeo FJ, Bautista OM, Esser MT, Sings HL, Nelson M, Boslego JW, Sattler C, Barr E, Paavonen J. Efficacy of a quadrivalent prophylactic human papillomavirus (types 6, 11, 16, and 18) L1 virus-like-particle vaccine against high-grade vulval and vaginal lesions: a combined analysis of three randomised clinical trials. Lancet. 2007 May 19;369(9574):1693-702. doi: 10.1016/S0140-6736(07)60777-6. PMID 17512854
- [Background] Perez G, Lazcano-Ponce E, Hernandez-Avila M, Garcia PJ, Munoz N, Villa LL, Bryan J, Taddeo FJ, Lu S, Esser MT, Vuocolo S, Sattler C, Barr E. Safety, immunogenicity, and efficacy of quadrivalent human papillomavirus (types 6, 11, 16, 18) L1 virus-like-particle vaccine in Latin American women. Int J Cancer. 2008 Mar 15;122(6):1311-8. doi: 10.1002/ijc.23260. PMID 18000825
- [Background] FUTURE II Study Group. Prophylactic efficacy of a quadrivalent human papillomavirus (HPV) vaccine in women with virological evidence of HPV infection. J Infect Dis. 2007 Nov 15;196(10):1438-46. doi: 10.1086/522864. Epub 2007 Oct 31. PMID 18008221
- [Background] Ault KA; Future II Study Group. Effect of prophylactic human papillomavirus L1 virus-like-particle vaccine on risk of cervical intraepithelial neoplasia grade 2, grade 3, and adenocarcinoma in situ: a combined analysis of four randomised clinical trials. Lancet. 2007 Jun 2;369(9576):1861-1868. doi: 10.1016/S0140-6736(07)60852-6. PMID 17544766
- [Background] Giuliano AR, Lazcano-Ponce E, Villa L, Nolan T, Marchant C, Radley D, Golm G, McCarroll K, Yu J, Esser MT, Vuocolo SC, Barr E. Impact of baseline covariates on the immunogenicity of a quadrivalent (types 6, 11, 16, and 18) human papillomavirus virus-like-particle vaccine. J Infect Dis. 2007 Oct 15;196(8):1153-62. doi: 10.1086/521679. Epub 2007 Sep 17. PMID 17955433
- [Background] Garland SM, Insinga RP, Sings HL, Haupt RM, Joura EA. Human papillomavirus infections and vulvar disease development. Cancer Epidemiol Biomarkers Prev. 2009 Jun;18(6):1777-84. doi: 10.1158/1055-9965.EPI-09-0067. PMID 19505910
- [Background] Skjeldestad FE, Mehta V, Sings HL, Ovreness T, Turpin J, Su L, Boerckel P, Roberts C, Bryan J, Jansen KU, Esser MT, Liaw KL. Seroprevalence and genital DNA prevalence of HPV types 6, 11, 16 and 18 in a cohort of young Norwegian women: study design and cohort characteristics. Acta Obstet Gynecol Scand. 2008;87(1):81-8. doi: 10.1080/00016340701714703. PMID 17943470
- [Background] Nygard M, Saah A, Munk C, Tryggvadottir L, Enerly E, Hortlund M, Sigurdardottir LG, Vuocolo S, Kjaer SK, Dillner J. Evaluation of the Long-Term Anti-Human Papillomavirus 6 (HPV6), 11, 16, and 18 Immune Responses Generated by the Quadrivalent HPV Vaccine. Clin Vaccine Immunol. 2015 Aug;22(8):943-8. doi: 10.1128/CVI.00133-15. Epub 2015 Jun 17. PMID 26084514
- [Background] Tay EH, Garland S, Tang G, Nolan T, Huang LM, Orloski L, Lu S, Barr E. Clinical trial experience with prophylactic HPV 6/11/16/18 VLP vaccine in young women from the Asia-Pacific region. Int J Gynaecol Obstet. 2008 Sep;102(3):275-83. doi: 10.1016/j.ijgo.2008.03.021. Epub 2008 Jun 16. PMID 18555997
- [Background] Majewski S, Bosch FX, Dillner J, Iversen OE, Kjaer SK, Munoz N, Olsson SE, Paavonen J, Sigurdsson K, Bryan J, Esser MT, Giacoletti K, James M, Taddeo F, Vuocolo S, Barr E. The impact of a quadrivalent human papillomavirus (types 6, 11, 16, 18) virus-like particle vaccine in European women aged 16 to 24. J Eur Acad Dermatol Venereol. 2009 Oct;23(10):1147-55. doi: 10.1111/j.1468-3083.2009.03266.x. Epub 2009 Apr 23. PMID 19453788
- [Background] Kjaer SK, Sigurdsson K, Iversen OE, Hernandez-Avila M, Wheeler CM, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Lehtinen M, Steben M, Bosch FX, Dillner J, Joura EA, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Maansson R, Lu S, Vuocolo S, Hesley TM, Saah A, Barr E, Haupt RM. A pooled analysis of continued prophylactic efficacy of quadrivalent human papillomavirus (Types 6/11/16/18) vaccine against high-grade cervical and external genital lesions. Cancer Prev Res (Phila). 2009 Oct;2(10):868-78. doi: 10.1158/1940-6207.CAPR-09-0031. Epub 2009 Sep 29. PMID 19789295
- [Background] FUTURE I/II Study Group; Dillner J, Kjaer SK, Wheeler CM, Sigurdsson K, Iversen OE, Hernandez-Avila M, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Lehtinen M, Steben M, Bosch FX, Joura EA, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan JT, Maansson R, Lu S, Vuocolo S, Hesley TM, Barr E, Haupt R. Four year efficacy of prophylactic human papillomavirus quadrivalent vaccine against low grade cervical, vulvar, and vaginal intraepithelial neoplasia and anogenital warts: randomised controlled trial. BMJ. 2010 Jul 20;341:c3493. doi: 10.1136/bmj.c3493. PMID 20647284
- [Background] Olsson SE, Kjaer SK, Sigurdsson K, Iversen OE, Hernandez-Avila M, Wheeler CM, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Tang GW, Ferris DG, Paavonen J, Lehtinen M, Steben M, Bosch FX, Dillner J, Joura EA, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Maansson R, Vuocolo S, Hesley TM, Saah A, Barr E, Haupt RM. Evaluation of quadrivalent HPV 6/11/16/18 vaccine efficacy against cervical and anogenital disease in subjects with serological evidence of prior vaccine type HPV infection. Hum Vaccin. 2009 Oct;5(10):696-704. doi: 10.4161/hv.5.10.9515. Epub 2009 Oct 1. PMID 19855170
- [Background] Haupt RM, Wheeler CM, Brown DR, Garland SM, Ferris DG, Paavonen JA, Lehtinen MO, Steben M, Joura EA, Giacoletti KE, Radley DR, James MK, Saah AJ, Sings HL; FUTURE I and II Investigators. Impact of an HPV6/11/16/18 L1 virus-like particle vaccine on progression to cervical intraepithelial neoplasia in seropositive women with HPV16/18 infection. Int J Cancer. 2011 Dec 1;129(11):2632-42. doi: 10.1002/ijc.25940. Epub 2011 Apr 13. PMID 21491420
- [Result] Kjaer SK, Nygard M, Dillner J, Brooke Marshall J, Radley D, Li M, Munk C, Hansen BT, Sigurdardottir LG, Hortlund M, Tryggvadottir L, Joshi A, Das R, Saah AJ. A 12-Year Follow-up on the Long-Term Effectiveness of the Quadrivalent Human Papillomavirus Vaccine in 4 Nordic Countries. Clin Infect Dis. 2018 Jan 18;66(3):339-345. doi: 10.1093/cid/cix797. PMID 29029053
- [Derived] Joura E, Kjaer SK, Bautista O, Luxembourg A, Saah A, Giuliano A. Effect of Prior 9-Valent Human Papillomavirus Vaccination on Subsequent Lower Genital Tract Dysplasia After Cervical Excisional Surgery. Obstet Gynecol. 2026 Jan 1;147(1):73-82. doi: 10.1097/AOG.0000000000006113. Epub 2025 Oct 30. PMID 41166720
- [Derived] Lehtinen M, Lagheden C, Luostarinen T, Eriksson T, Apter D, Bly A, Gray P, Harjula K, Heikkila K, Hokkanen M, Karttunen H, Kuortti M, Nieminen P, Nummela M, Paavonen J, Palmroth J, Petaja T, Pukkala E, Soderlund-Strand A, Veivo U, Dillner J. Human papillomavirus vaccine efficacy against invasive, HPV-positive cancers: population-based follow-up of a cluster-randomised trial. BMJ Open. 2021 Dec 30;11(12):e050669. doi: 10.1136/bmjopen-2021-050669. PMID 35149535
- [Derived] Enerly E, Berger S, Kjaer SK, Sundstrom K, Campbell S, Tryggvadottir L, Munk C, Hortlund M; Thomas Group. Electronic address: thomas_group@merck.com; Joshi A, Saah AJ, Nygard M. Use of real-world data for HPV vaccine trial follow-up in the Nordic region. Contemp Clin Trials. 2020 May;92:105996. doi: 10.1016/j.cct.2020.105996. Epub 2020 Apr 1. PMID 32247041
- [Derived] Doshi P, Bourgeois F, Hong K, Jones M, Lee H, Shamseer L, Spence O, Jefferson T. Adjuvant-containing control arms in pivotal quadrivalent human papillomavirus vaccine trials: restoration of previously unpublished methodology. BMJ Evid Based Med. 2020 Dec;25(6):213-219. doi: 10.1136/bmjebm-2019-111331. Epub 2020 Mar 17. PMID 32184277
- [Derived] Giuliano AR, Joura EA, Garland SM, Huh WK, Iversen OE, Kjaer SK, Ferenczy A, Kurman RJ, Ronnett BM, Stoler MH, Bautista OM, Moeller E, Ritter M, Shields C, Luxembourg A. Nine-valent HPV vaccine efficacy against related diseases and definitive therapy: comparison with historic placebo population. Gynecol Oncol. 2019 Jul;154(1):110-117. doi: 10.1016/j.ygyno.2019.03.253. Epub 2019 Apr 11. PMID 30982556
- [Derived] Garland SM, Joura EA, Ault KA, Bosch FX, Brown DR, Castellsague X, Ferenczy A, Ferris DG, Giuliano AR, Hernandez-Avila M, Huh WK, Iversen OE, Kjaer SK, Kurman RJ, Luna J, Monsonego J, Munoz N, Paavonen J, Pitisuttihum P, Ronnett BM, Steben M, Stoler MH, Wheeler CM, Wiley DJ, Perez G, Saah AJ, Luxembourg A, Li S, DiNubile MJ, Wagner M, Velicer C. Human Papillomavirus Genotypes From Vaginal and Vulvar Intraepithelial Neoplasia in Females 15-26 Years of Age. Obstet Gynecol. 2018 Aug;132(2):261-270. doi: 10.1097/AOG.0000000000002736. PMID 29995724
- [Derived] Castellsague X, Ault KA, Bosch FX, Brown D, Cuzick J, Ferris DG, Joura EA, Garland SM, Giuliano AR, Hernandez-Avila M, Huh W, Iversen OE, Kjaer SK, Luna J, Monsonego J, Munoz N, Myers E, Paavonen J, Pitisuttihum P, Steben M, Wheeler CM, Perez G, Saah A, Luxembourg A, Sings HL, Velicer C. Human papillomavirus detection in cervical neoplasia attributed to 12 high-risk human papillomavirus genotypes by region. Papillomavirus Res. 2016 Dec;2:61-69. doi: 10.1016/j.pvr.2016.03.002. Epub 2016 Mar 14. PMID 29074187
- [Derived] Clark LR, Myers ER, Huh W, Joura EA, Paavonen J, Perez G, James MK, Sings HL, Haupt RM, Saah AJ, Garner EI. Clinical trial experience with prophylactic human papillomavirus 6/11/16/18 vaccine in young black women. J Adolesc Health. 2013 Mar;52(3):322-9. doi: 10.1016/j.jadohealth.2012.07.003. Epub 2012 Aug 15. PMID 23299013
- [Derived] Ruiz AM, Ruiz JE, Gavilanes AV, Eriksson T, Lehtinen M, Perez G, Sings HL, James MK, Haupt RM; FUTURE I and II Study Group. Proximity of first sexual intercourse to menarche and risk of high-grade cervical disease. J Infect Dis. 2012 Dec 15;206(12):1887-96. doi: 10.1093/infdis/jis612. Epub 2012 Oct 12. PMID 23066159
- [Derived] Joura EA, Garland SM, Paavonen J, Ferris DG, Perez G, Ault KA, Huh WK, Sings HL, James MK, Haupt RM; FUTURE I and II Study Group. Effect of the human papillomavirus (HPV) quadrivalent vaccine in a subgroup of women with cervical and vulvar disease: retrospective pooled analysis of trial data. BMJ. 2012 Mar 27;344:e1401. doi: 10.1136/bmj.e1401. PMID 22454089
- [Derived] Lehtinen M, Ault KA, Lyytikainen E, Dillner J, Garland SM, Ferris DG, Koutsky LA, Sings HL, Lu S, Haupt RM, Paavonen J; FUTURE I and II Study Group. Chlamydia trachomatis infection and risk of cervical intraepithelial neoplasia. Sex Transm Infect. 2011 Aug;87(5):372-6. doi: 10.1136/sti.2010.044354. Epub 2011 Apr 6. PMID 21471141
- [Derived] Ault KA, Joura EA, Kjaer SK, Iversen OE, Wheeler CM, Perez G, Brown DR, Koutsky LA, Garland SM, Olsson SE, Tang GW, Ferris DG, Paavonen J, Steben M, Bosch FX, Majewski S, Munoz N, Sings HL, Harkins K, Rutkowski MA, Haupt RM, Garner EI; FUTURE I and II Study Group. Adenocarcinoma in situ and associated human papillomavirus type distribution observed in two clinical trials of a quadrivalent human papillomavirus vaccine. Int J Cancer. 2011 Mar 15;128(6):1344-53. doi: 10.1002/ijc.25723. Epub 2011 Jan 12. PMID 20949623
- [Derived] Garland SM, Ault KA, Gall SA, Paavonen J, Sings HL, Ciprero KL, Saah A, Marino D, Ryan D, Radley D, Zhou H, Haupt RM, Garner EIO; Quadrivalent Human Papillomavirus Vaccine Phase III Investigators. Pregnancy and infant outcomes in the clinical trials of a human papillomavirus type 6/11/16/18 vaccine: a combined analysis of five randomized controlled trials. Obstet Gynecol. 2009 Dec;114(6):1179-1188. doi: 10.1097/AOG.0b013e3181c2ca21. PMID 19935017
- [Derived] Brown DR, Kjaer SK, Sigurdsson K, Iversen OE, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Steben M, Bosch FX, Dillner J, Joura EA, Kurman RJ, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Lupinacci LC, Giacoletti KE, Sings HL, James M, Hesley TM, Barr E. The impact of quadrivalent human papillomavirus (HPV; types 6, 11, 16, and 18) L1 virus-like particle vaccine on infection and disease due to oncogenic nonvaccine HPV types in generally HPV-naive women aged 16-26 years. J Infect Dis. 2009 Apr 1;199(7):926-35. doi: 10.1086/597307. PMID 19236279
- [Derived] Wheeler CM, Kjaer SK, Sigurdsson K, Iversen OE, Hernandez-Avila M, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Steben M, Bosch FX, Dillner J, Joura EA, Kurman RJ, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Lupinacci LC, Giacoletti KE, James M, Vuocolo S, Hesley TM, Barr E. The impact of quadrivalent human papillomavirus (HPV; types 6, 11, 16, and 18) L1 virus-like particle vaccine on infection and disease due to oncogenic nonvaccine HPV types in sexually active women aged 16-26 years. J Infect Dis. 2009 Apr 1;199(7):936-44. doi: 10.1086/597309. PMID 19236277
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female participants were randomized to receive quadrivalent human papillomavirus (qHPV) vaccine (GARDASIL™) or placebo in the Base Study (V501-015, NCT00092534), and were followed for 4 years. Participants who received placebo in the Base Study were eligible to receive the 3-dose qHPV vaccine series during the Base Study Extension (EXT).
Pre-assignment Details: Participants who received 3 doses of qHPV vaccine either during the Base Study or Base Study EXT were eligible for enrollment in the Long-Term Follow-Up (LTFU) Study (V501-015-21).
  The 10-year-long registry-based LTFU was conducted at 4 National Registry Study Centers (NRSC) in Denmark, Iceland, Norway, and Sweden.
Groups:
- Base Study Group 1: qHPV Vaccine: During the Base Study, participants received 3 qHPV vaccinations (at Day 1, Month 2 and Month 6) and were followed for up to 4 years.
- Base Study Group 2: Placebo: During the Base Study, participants received 3 placebo vaccinations (at Day 1, Month 2 and Month 6) and were followed for up to 4 years.
- Base Study EXT: Participants who received placebo (N=581) or an incomplete qHPV vaccine regimen (N=13) were enrolled to receive qHPV vaccine during the base study extension; participants designated as "Not Completed" are those who did not complete all three vaccinations and/or all required follow-up visits.
- LTFU: Cohort 1: Participants who received qHPV vaccine in the Base Study with approximately 4 years of follow-up in the Base Study and 10 years of follow-up in the LTFU. Cohort 1 provided a total of approximately 14 years of follow-up post-vaccination.
- LTFU: Cohort 2: Participants who received placebo in the Base Study and qHPV vaccine after completion of the Base Study and prior to entry into the LTFU. Cohort 2 provided a total of approximately 10 years of follow-up post-vaccination.
Period: Base Study Vaccination Period
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo | Base Study EXT | LTFU: Cohort 1 | LTFU: Cohort 2
Started | 6087 | 6080 | 0 | 0 | 0
Completed | 5916 | 5954 | 0 | 0 | 0
Not Completed | 171 | 126 | 0 | 0 | 0
Not completed — Randomized not Vaccinated | 5 | 5 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 0 | 0 | 0
Not completed — Death | 5 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 41 | 37 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 9 | 7 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 85 | 58 | 0 | 0 | 0
Not completed — Moved | 14 | 12 | 0 | 0 | 0
Not completed — New Medical History (Not AEs) | 5 | 0 | 0 | 0 | 0
Not completed — Travel | 1 | 0 | 0 | 0 | 0
Not completed — Site Closed | 0 | 1 | 0 | 0 | 0
Period: Base Study Follow-Up Period
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo | Base Study EXT | LTFU: Cohort 1 | LTFU: Cohort 2
Started | 5942 (Includes subjects who did not receive 3 doses of vaccine/placebo but continued into the follow-up.) | 5971 (Includes subjects who did not receive 3 doses of vaccine/placebo but continued into the follow-up.) | 0 | 0 | 0
Completed | 5626 | 5277 | 0 | 0 | 0
Not Completed | 316 | 694 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 120 | 146 | 0 | 0 | 0
Not completed — Pregnancy | 6 | 10 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 71 | 62 | 0 | 0 | 0
Not completed — Moved | 62 | 58 | 0 | 0 | 0
Not completed — Travel | 10 | 7 | 0 | 0 | 0
Not completed — Site Closed | 0 | 2 | 0 | 0 | 0
Not completed — Subjects continuing | 27 | 31 | 0 | 0 | 0
Not completed — Subjects in extension | 15 | 371 | 0 | 0 | 0
Period: Base Study EXT
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo | Base Study EXT | LTFU: Cohort 1 | LTFU: Cohort 2
Started | 0 | 0 | 594 | 0 | 0
Completed | 0 | 0 | 449 | 0 | 0
Not Completed | 0 | 0 | 145 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 41 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 18 | 0 | 0
Not completed — Participant moved | 0 | 0 | 6 | 0 | 0
Not completed — Travel | 0 | 0 | 2 | 0 | 0
Not completed — Site closed | 0 | 0 | 21 | 0 | 0
Not completed — Study ended | 0 | 0 | 29 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 15 | 0 | 0
Period: Long-Term Follow-Up (LTFU) Study
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo | Base Study EXT | LTFU: Cohort 1 | LTFU: Cohort 2
Started (Eligible for inclusion in the LTFU study) | 0 | 0 | 0 | 2750 (Some Base Study participants did not consent for inclusion in the LTFU.) | 2097 (Some Base Study participants did not consent for inclusion in the LTFU.)
Started: Registry-based Effectiveness (Eligible and consented to inclusion in registry-based searches for effectiveness information) | 0 | 0 | 0 | 2650 | 2050
Started: Immunogenicity Analysis (Eligible and consented to provide blood samples for immunogenicity anaysis) | 0 | 0 | 0 | 2385 | 1849
Started: Registry-based Safety (Eligible and consented to inclusion in registry-based searches for safety information) | 0 | 0 | 0 | 2448 | 1888
Completed | 0 | 0 | 0 | 2749 | 2097
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis population is from the V501-015 Base Study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo | Total
Number analyzed (Participants) | 6087 | 6080 | 12167
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (2.2) | 19.9 (2.1) | 19.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6087 | 6080 | 12167
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 151 | 135 | 286
  Black | 171 | 227 | 398
  Hispanic American | 555 | 557 | 1112
  Native American | 1 | 1 | 2
  White | 4584 | 4550 | 9134
  Other-Unspecified | 625 | 610 | 1235

OUTCOME MEASURES:

1. Primary Outcome: Incidence of the Composite Endpoint of Human Papillomavirus (HPV) 16/18-related Cervical Intraepithelial Neoplasia (CIN) 2 or Worse in the Base Study
Description: This measure is defined to have occurred when, on a single cervical biopsy, endocervical curettage (ECC), loop electrosurgical excision procedure (LEEP), or conization specimen, there was HPV Vaccine consensus diagnosis of CIN 2 or worse up to 4 years after the first vaccination. For this measure, CIN 2 or worse includes CIN 2, CIN 3, adenocarcinoma in situ (AIS) or cervical cancer related to HPV 16 or 18.
Time Frame: Up to 4 years
Population: Participants who received 3 qHPV doses in 1 year, had no protocol violations that could affect evaluation of vaccine efficacy, were polymerase chain reaction (PCR)-negative and seronegative based on competitive Luminex immunoassay (cLIA) to the relevant type at Day 1 and PCR-negative to the relevant type through Month 7, and had data available.
Measure: Number; unit: Incidence per 100 person-years
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo
Number analyzed (Participants) | 5306 | 5262
Incidence per 100 person-years | 0.0 | 0.4
Statistical Analysis 1: Comparison: Base Study Group 1: qHPV Vaccine vs Base Study Group 2: Placebo; Test type: Superiority or Other; Percent relative risk reduction = 96.6, 95% CI [88.2 to 99.6] — Confidence Interval (CI) based on binomial tail probabilities and not from a dispersion parameter

2. Primary Outcome: Incidence of the Composite Endpoint of Human Papillomavirus (HPV) 16/18-related Cervical Intraepithelial Neoplasia (CIN) 2 or Worse in the Long-term Follow-up (LTFU) Study
Description: This measure is defined to have occurred when, on a single cervical biopsy, endocervical curettage (ECC), loop electrosurgical excision procedure (LEEP), or conization specimen, there was HPV Vaccine Nordic pathology panel (NPP) consensus diagnosis of CIN 2 or worse up to 14 years after the first vaccination. For this measure, CIN 2 or worse includes CIN 2, CIN 3, AIS or cervical cancer related to HPV 16 or 18. Only participants who received qHPV vaccine during the Base Study vaccination period and consented for inclusion in the LTFU are included. Because the objective was to demonstrate qHPV vaccine prophylactic efficacy at 14 years, Cohort 2 was not included in the analysis.
Time Frame: Up to 14 years since Vaccine Dose 1
Population: Participants in Cohort 1 who received 3 qHPV vaccine doses in 1 year, had no protocol violations that could affect evaluation of efficacy, had been PCR-negative and seronegative based on cLIA at Day 1 and PCR-negative through Month 7 of the Base Study to the relevant HPV type(s), and had LTFU data available.
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2121
Incidence per 100 person-years | 0.0 [0.0 to 0.1]

3. Primary Outcome: Incidence of the Composite Endpoint of HPV16/18-related CIN 2 or Worse in the Long-term Follow-up (LTFU) Study
Description: This measure is defined to have occurred when, on a single cervical biopsy, ECC, LEEP, or conization specimen, there was HPV Vaccine NPP consensus diagnosis of CIN 2 or worse up to 22 years after the first vaccination. For this measure, CIN 2 or worse includes CIN 2, CIN 3, AIS or cervical cancer related to HPV 16 or 18. Only participants who received qHPV vaccine during the Base Study vaccination period and consented for inclusion in the LTFU will be included.
Time Frame: up to 22 years post Vaccination Dose 1
Reporting Status: Not Posted, anticipated posting 2026-11

4. Secondary Outcome: Number of Participants With Anti-Human Papillomavirus (HPV) 6 Titer ≥20 mMU/mL Based on Competitive Luminex Immunoassay (cLIA) in the Base Study
Description: Anti-HPV levels >20 mMU/mL neutralize a large input load of HPV 6 pseudovirions in vitro; thus, the number of participants with anti-HPV 6 ≥20 mMU/mL 4 four weeks after the third quadrivalent HPV (qHPV) or placebo vaccination in the Base Study was determined.
Time Frame: Month 7 (4 weeks after Vaccination 3)
Population: Participants who received 3 qHPV vaccine doses and had Month 7 results within acceptable ranges, had no protocol violations that could affect evaluation of vaccine immunogenicity, and were polymerase chain reaction (PCR)-negative and seronegative based on cLIA to the relevant type at Day 1 and PCR-negative to the relevant type through Month 7.
Measure: Number; unit: Number of Participants
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo
Number analyzed (Participants) | 1056 | 1057
Number of Participants | 1054 | 13

5. Secondary Outcome: Number of Participants With Anti-Human Papillomavirus (HPV) 11 Titer ≥16 mMU/mL Based on Competitive Luminex Immunoassay (cLIA) in the Base Study
Description: Anti-HPV levels >20 mMU/mL neutralize a large input load of HPV 11 virions in vitro; thus, the number of participants with anti-HPV 11 ≥16 mMU/mL 4 four weeks after the third quadrivalent HPV (qHPV) or placebo vaccination in the Base Study was determined.
Time Frame: Week 4 Postdose 3
Population: as for outcome 4
Measure: Number; unit: Number of Participants
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo
Number analyzed (Participants) | 1057 | 1057
Number of Participants | 1054 | 5

6. Secondary Outcome: Number of Participants With Anti-Human Papillomavirus (HPV) 16 Titer ≥20 mMU/mL Based on Competitive Luminex Immunoassay (cLIA) in the Base Study
Description: Anti-HPV levels >20 mMU/mL neutralize a large input load of HPV 16 pseudovirions in vitro; thus, the number of participants with anti-HPV 16 ≥20 mMU/mL 4 four weeks after the third quadrivalent HPV (qHPV) or placebo vaccination in the Base Study was determined.
Time Frame: Week 4 Postdose 3
Population: as for outcome 4
Measure: Number; unit: Number of Participants
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo
Number analyzed (Participants) | 1017 | 994
Number of Participants | 1014 | 15

7. Secondary Outcome: Number of Participants With Anti-Human Papillomavirus (HPV) 18 Titer ≥24 mMU/mL Based on Competitive Luminex Immunoassay (cLIA) in the Base Study
Description: Anti-HPV levels >20 mMU/mL neutralize a large input load of HPV 18 pseudovirions in vitro; thus, the number of participants with anti-HPV 18 ≥24 mMU/mL 4 four weeks after the third quadrivalent HPV (qHPV) or placebo vaccination in the Base Study was determined.
Time Frame: Week 4 Postdose 3
Population: as for outcome 4
Measure: Number; unit: Number of Participants
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo
Number analyzed (Participants) | 1140 | 1119
Number of Participants | 1133 | 12

8. Secondary Outcome: Incidence of the Composite Endpoint of Human Papillomavirus (HPV) 31/33/35/39/45/51/52/56/58/59-related Cervical Intraepithelial Neoplasia (CIN) Grade 2 or Worse in the Long-term Follow-up (LTFU) Study
Description: This measure is defined to have occurred when, on a single cervical biopsy, endocervical curettage (ECC), loop electrosurgical excision procedure (LEEP), or conization specimen, there was HPV Vaccine Nordic pathology panel (NPP) consensus diagnosis of CIN 2 or worse related to nonvaccine HPV types up to 14 years after the first vaccination. For this measure, CIN 2 or worse includes CIN 2, CIN 3, AIS or cervical cancer related to nonvaccine HPV types 31, 33, 35, 39, 45, 51, 52, 56, 58, or 59. Only participants who received qHPV vaccine during the Base Study vaccination period and consented for inclusion in the LTFU are included. Because the objective was to demonstrate qHPV vaccine prophylactic efficacy at 14 years, Cohort 2 was not included in the analysis.
Time Frame: Up to 14 years since Vaccination Dose 1
Population: Participants in Cohort 1 who had received ≥1 qHPV vaccination, had any follow up visit in the LTFU, and had been PCR-negative and seronegative based on cLIA to the appropriate HPV type(s) at Day 1.
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2355
Incidence per 100 person-years | 0.2 [0.1 to 0.2]

9. Secondary Outcome: Incidence of the Composite Endpoint of HPV 6/11/16/18-related CIN (Any Grade), AIS, Cervical Cancer, Vulvar Cancer or Vaginal Cancer the Long-term Follow-up (LTFU) Study
Description: This measure was defined to have occurred if on a single biopsy or excised tissue, there was the NPP consensus diagnosis of CIN 1, CIN 2, CIN 3, AIS, cervical cancer, vulvar cancer or vaginal cancer AND at least 1 of HPV types 6, 11, 16 or 18 was detected by Thin-section PCR in an adjacent section from the same tissue block. Only participants who received qHPV vaccine during the Base Study vaccination period and consented for inclusion in the LTFU are included. Because the objective was to demonstrate qHPV vaccine prophylactic efficacy at 14 years, Cohort 2 was not included in the analysis.
Time Frame: Up to 14 years since Vaccination Dose 1
Population: Participants in Cohort 1 who received 3 qHPV vaccine doses in 1 year, had no protocol violations that could affect efficacy, had been PCR-negative and seronegative based on cLIA at Day 1 and PCR-negative through Month 7 of the Base Study to relevant HPV type(s), and had LTFU data available.
Measure: Number (95% Confidence Interval); unit: Incidence per 100 person-years
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2312
Incidence per 100 person-years | 0.1 [0.1 to 0.1]

10. Secondary Outcome: Incidence of the Composite Endpoint of HPV 6/11/16/18-related CIN (Any Grade), AIS, Cervical Cancer, Vulvar Cancer or Vaginal Cancer the Long-term Follow-up (LTFU) Study
Description: This measure is defined to have occurred if on a single biopsy or excised tissue, there is the NPP consensus diagnosis of CIN 1, CIN 2, CIN 3, AIS, cervical cancer, vulvar cancer or vaginal cancer AND at least 1 of HPV types 6, 11, 16 or 18 is detected by Thin-section PCR in an adjacent section from the same tissue block.
Time Frame: up to 22 years since Vaccination Dose 1
Reporting Status: Not Posted, anticipated posting 2026-11

11. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV Types 6, 11, 16, and 18 at Month 108 Assessed by Competitive Luminex Immunoassay (cLIA) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to human papillomavirus (HPV) types were measured using cLIA. Because the objective was to demonstrate antibody persistence at 14 years following vaccination in susceptible individuals, Cohort 2 was not included in the analysis.
Time Frame: At 108 months since Vaccination Dose 1
Population: Participants in Cohort 1 who received 3 qHPV vaccine doses in 1 year, had no protocol violations that could affect evaluation of vaccine immunogenicity, and were PCR-negative and seronegative based on cLIA to relevant type at Day 1 and PCR-negative to the relevant type through Month 7. No data were collected for Cohort 2.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2750
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 1234
  Anti-HPV 6 | 89.2 [84.7 to 94.0]
  Anti-HPV 11: number analyzed (Participants) | 1234
  Anti-HPV 11 | 85.2 [80.7 to 90.0]
  Anti-HPV 16: number analyzed (Participants) | 1179
  Anti-HPV 16 | 348.6 [328.3 to 370.2]
  Anti-HPV 18: number analyzed (Participants) | 1332
  Anti-HPV 18 | 32.5 [30.2 to 34.9]

12. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV Types 6, 11, 16, and 18 at Month 168 Assessed by Competitive Luminex Immunoassay (cLIA) in the Long-Term Follow-Up (LTFU) Study
Description: as for outcome 11
Time Frame: At 168 months since Vaccination Dose 1
Population: Participants in Cohort 1 who received 3 qHPV vaccine doses within 1 year, had no protocol violations that could affect evaluation of vaccine immunogenicity, and were PCR-negative and seronegative based on cLIA to the relevant type at Day 1 and PCR-negative to the relevant type through Month 7.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2750
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 1058
  Anti-HPV 6 | 78.4 [73.8 to 83.2]
  Anti-HPV 11: number analyzed (Participants) | 1058
  Anti-HPV 11 | 66.8 [62.6 to 71.3]
  Anti-HPV 16: number analyzed (Participants) | 1005
  Anti-HPV 16 | 291.2 [272.1 to 311.5]
  Anti-HPV 18: number analyzed (Participants) | 1131
  Anti-HPV 18 | 26.1 [24.1 to 28.2]

13. Secondary Outcome: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 108 Assessed by Competitive Luminex Immunoassay (cLIA) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to human papillomavirus (HPV) types were measured using cLIA. Seropositivity was assessed by competitive Luminex Immunoassay (cLIA); the serostatus cut-offs for anti-HPV 6, 11, 16 and 18 serum cLIA were 20, 16, 20 and 24 milliMerck units (mMU)/mL, respectively. Because the objective was to demonstrate antibody persistence at 14 years following vaccination in susceptible individuals, Cohort 2 was not included in the analysis.
Time Frame: At 108 months since Vaccination Dose 1
Population: Participants in Cohort 1 who received 3 qHPV vaccine doses within 1 year, had no protocol violations that could affect evaluation of vaccine immunogenicity, and were PCR-negative and seronegative based on cLIA to the relevant type at Day 1 and PCR-negative to the relevant type through Month 7. No data were collected for Cohort 2.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2750
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 1234
  Anti-HPV 6 | 94.4 [93.0 to 95.6]
  Anti-HPV 11: number analyzed (Participants) | 1234
  Anti-HPV 11 | 95.5 [94.1 to 96.6]
  Anti-HPV 16: number analyzed (Participants) | 1179
  Anti-HPV 16 | 99.1 [98.3 to 99.5]
  Anti-HPV 18: number analyzed (Participants) | 1332
  Anti-HPV 18 | 59.9 [57.2 to 62.6]

14. Secondary Outcome: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 168 Assessed by Competitive Luminex Immunoassay (cLIA) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to human papillomavirus (HPV) types were measured using cLIA. Seropositivity was assessed by cLIA; the serostatus cut-offs for anti-HPV 6, 11, 16 and 18 serum cLIA were 20, 16, 20 and 24 milliMerck units (mMU)/mL, respectively. Because the objective was to demonstrate antibody persistence at 14 years following vaccination in susceptible individuals, Cohort 2 was not included in the analysis.
Time Frame: At 168 months since Vaccination Dose 1
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2750
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 1058
  Anti-HPV 6 | 90.6 [88.7 to 92.3]
  Anti-HPV 11: number analyzed (Participants) | 1058
  Anti-HPV 11 | 91.1 [89.2 to 92.8]
  Anti-HPV 16: number analyzed (Participants) | 1005
  Anti-HPV 16 | 98.3 [97.3 to 99.0]
  Anti-HPV 18: number analyzed (Participants) | 1131
  Anti-HPV 18 | 52.4 [49.5 to 55.4]

15. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV Types 6, 11, 16, and 18 at Month 108 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to human papillomavirus (HPV) types were measured using IgG LIA. Because the objective was to demonstrate antibody persistence at 14 years following vaccination in susceptible individuals, Cohort 2 was not included in the analysis.
Time Frame: At 108 months since Vaccination Dose 1
Population: Participants in Cohort 1 who received 3 qHPV vaccine doses within 1 year, had no protocol violations that could affect evaluation of vaccine immunogenicity, were PCR-negative and seronegative based on cLIA to the relevant type at Day 1 and PCR-negative to the relevant type through Month 7. No data were collected for Cohort 2.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2750
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 1235
  Anti-HPV 6 | 95.2 [90.5 to 100.1]
  Anti-HPV 11: number analyzed (Participants) | 1235
  Anti-HPV 11 | 67.4 [64.3 to 70.8]
  Anti-HPV 16: number analyzed (Participants) | 1181
  Anti-HPV 16 | 346.1 [327.3 to 365.9]
  Anti-HPV 18: number analyzed (Participants) | 1333
  Anti-HPV 18 | 46.1 [43.3 to 49.2]

16. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV Types 6, 11, 16, and 18 at Month 168 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA) in the Long-Term Follow-Up (LTFU) Study
Description: as for outcome 15
Time Frame: At 168 months since Vaccination Dose 1
Population: Participants in Cohort 1 who received 3 qHPV vaccine doses within 1 year, had no protocol violations that could affect evaluation of vaccine immunogenicity, were PCR-negative and seronegative based on cLIA to the relevant type at Day 1 and PCR-negative to the relevant type through Month 7.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2750
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 1054
  Anti-HPV 6 | 81.2 [76.1 to 86.5]
  Anti-HPV 11: number analyzed (Participants) | 1055
  Anti-HPV 11 | 53.5 [50.2 to 57.0]
  Anti-HPV 16: number analyzed (Participants) | 1000
  Anti-HPV 16 | 290.2 [271.0 to 310.8]
  Anti-HPV 18310.8: number analyzed (Participants) | 1036
  Anti-HPV 18310.8 | 36.5 [33.7 to 39.5]

17. Secondary Outcome: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 108 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to HPV types were measured using anti-HPV IgG LIA. The serostatus cut-offs for IgG LIA anti-HPV 6, 11, 16 and 18 at Month 108 were 15, 15, 7, and 10 milliMerck units (mMU)/mL, respectively. Because the objective was to demonstrate antibody persistence at 14 years following vaccination in susceptible individuals, Cohort 2 was not included in the analysis.
Time Frame: At 108 months since Vaccination Dose 1
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2750
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 1235
  Anti-HPV 6 | 97.6 [96.6 to 98.4]
  Anti-HPV 11: number analyzed (Participants) | 1235
  Anti-HPV 11 | 96.3 [95.1 to 97.3]
  Anti-HPV 16: number analyzed (Participants) | 1181
  Anti-HPV 16 | 100.0 [99.7 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 1333
  Anti-HPV 18 | 91.4 [89.7 to 92.8]

18. Secondary Outcome: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 168 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to HPV types were measured using anti-HPV IgG LIA. The serostatus cut-offs for IgG LIA anti-HPV 6, 11, 16 and 18 at Month 168 were 9, 6, 5, and 5 milliMerck units (mMU)/mL, respectively. Because the objective was to demonstrate antibody persistence at 14 years following vaccination in susceptible individuals, Cohort 2 was not included in the analysis.
Time Frame: At 168 months since Vaccination Dose 1
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | LTFU: Cohort 1
Number analyzed (Participants) | 2750
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 1054
  Anti-HPV 6 | 98.1 [97.1 to 98.8]
  Anti-HPV 11: number analyzed (Participants) | 1055
  Anti-HPV 11 | 98.0 [97.0 to 98.8]
  Anti-HPV 16: number analyzed (Participants) | 1000
  Anti-HPV 16 | 100.0 [99.6 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 1036
  Anti-HPV 18 | 93.8 [92.2 to 95.2]

19. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV Types 6, 11, 16, and 18 at Month 216 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to human papillomavirus (HPV) types will be measured using IgG LIA..
Time Frame: At 216 months since Vaccination Dose 1
Reporting Status: Not Posted, anticipated posting 2026-11

20. Secondary Outcome: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 216 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA) ) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to HPV types will be measured using anti-HPV IgG LIA. The serostatus cut-offs for IgG LIA anti-HPV 6, 11, 16 and 18 are 15, 15, 7, and 10 milliMerck units (mMU)/mL, respectively. The percentage of participants that are seropositive for each type will be summarized.
Time Frame: At 216 months since Vaccination Dose 1
Reporting Status: Not Posted, anticipated posting 2026-11

21. Secondary Outcome: Geometric Mean Titers (GMTs) to HPV Types 6, 11, 16, and 18 at Month 264 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA) in the Long-Term Follow-Up (LTFU) Study
Description: Antibodies to human papillomavirus (HPV) types will be measured using IgG LIA..
Time Frame: At 264 months since Vaccination Dose 1
Reporting Status: Not Posted, anticipated posting 2026-11

22. Secondary Outcome: Percentage of Participants With Seropositivity to HPV Types 6, 11, 16, and 18 at Month 264 Assessed by Immunoglobulin G Luminex Immunoassay (IgG LIA) in the Long-Term Follow-Up (LTFU) Study
Description: as for outcome 20
Time Frame: At 264 months since Vaccination Dose 1
Reporting Status: Not Posted, anticipated posting 2026-11

ADVERSE EVENTS:
Time Frame: From randomization in the Base Study to up to 10 years after completion of the Base Study (up to 14 years)
Description: The number of participants at risk includes randomized participants who had follow-up data available. Both serious adverse events (SAEs) and nonserious AEs were collected in the Base Study. Safety data for the LTFU were evaluated based on health outcomes data available from the national registries; in addition, AEs and SAEs associated with blood draws at LTFU Year 5 and Year 10 were also collected.
Groups:
- Base Study Group 1: qHPV Vaccine: During the Base Study, participants received 3 qHPV vaccinations (at Day 1, Month 2 and Month 6) during the Vaccination Period and were followed for up to 4 years during the Base Study Follow-Up.
- Base Study Group 2: Placebo: Participants received 3 placebo vaccinations (at Day 1, Month 2 and Month 6) during the Base Study Vaccination Period, and then received 3 qHPV vaccinations during the 4-year Base Study EXT.
- LTFU: Cohort 2: Participants who received placebo in the Base Study and qHPV vaccine after completion of the Base Study and prior to entry into the LTFU. Cohort 2 provided a total of approximately 10 years of follow-up post-vaccination in the LTFU.
Arm/Group | Base Study Group 1: qHPV Vaccine | Base Study Group 2: Placebo | Base Study EXT | LTFU: Cohort 1 | LTFU: Cohort 2
All-Cause Mortality (participants affected / at risk) | 7/6082 | 5/6075 | 0/594 | 2/2448 | 1/1888
Serious Adverse Events (participants affected / at risk) | 46/6082 | 56/6075 | 1/594 | 0/2448 | 0/1888
Other Adverse Events (participants affected / at risk) | 551/6082 | 499/6075 | 0/594 | 0/2448 | 0/1888
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Base Study Group 1: qHPV Vaccine (N=6082) | Base Study Group 2: Placebo (N=6075) | Base Study EXT (N=594) | LTFU: Cohort 1 (N=2448) | LTFU: Cohort 2 (N=1888)
Appendicitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Endometritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infective thrombosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pelvic Inflammatory disease (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Typhoid fever (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Uterine infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Failed forceps delivery (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 3 | 4 | 0 | 0 | 0
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Brow presentation (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 5 | 0 | 0 | 0
Cervix dystocia (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0
Failed trial of labour (Pregnancy, puerperium and perinatal conditions) | 3 | 3 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 3 | 2 | 0 | 0 | 0
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 3 | 5 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1/6021 | 0/6033 | 0 | 0/594 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Hypersensitivty (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0
Vaginal laceration (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0
Injection site joint movement impairment (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Base Study Group 1: qHPV Vaccine (N=6082) | Base Study Group 2: Placebo (N=6075) | Base Study EXT (N=594) | LTFU: Cohort 1 (N=2448) | LTFU: Cohort 2 (N=1888)
Injection site erythema (General disorders) | 142 | 120 | 0 | 0 | 0
Injection site pain (General disorders) | 503 | 433 | 0 | 0 | 0
Injection site swelling (General disorders) | 97 | 76 | 0 | 0 | 0
Headache (Nervous system disorders) | 162 | 167 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.